CLINICAL TRIAL: NCT05361460
Title: Patients Experiences of Early Postoperative Cognition and Its Relation to Cognitive Decline and Inflammatory Responses: a Mixed Methods Study
Brief Title: Patients Experiences of Early Postoperative Cognition
Acronym: COME
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ulrica Nilsson, Professor, Karolinska Institutet
Other Study IDs: 2019-02968
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Cognitive Decline; Biomarkers; Postoperative Recovery; Joint Replacement Surgery
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing major elective joint replacement surgery: patients ≥60 years that are undergoing major elective joint replacement surgery Exclusion criteria: a score on the mini-mental state examination (MMSE) at screening of ≤ 22 i.e. suspected dementia; < 60 years of age; suffering from a nervous system disease; taking tranquillisers or antidepressants; underwent a surgical procedure in the previous six months; or inability to read and speak Swedish; suffering from a severe visual or auditory disorder, alcoholism or drug dependence
  Interventions: Other: Cognitive decline

INTERVENTIONS:
Other: Cognitive decline — This is an observation study with the aim of explore patients' experiences of their early and late postoperative cognition after major orthopaedic surgery in relation to postoperative cognitive function assessed with validated neuropsychological tests, inflammatory signalling molecules and quality of postoperative recovery as well as to describe the relative's view of early postoperative cognition.

SUMMARY:
The study has a mixed-methods design i.e. integration of qualitative and quantitative data within a single investigation. Participants included will be patients ≥60 years that are undergoing major elective joint replacement surgery (n=40) and their relative. Patient's experience of his/her cognition will be capture by interviews on postoperative day 13-16 during the follow-up visit and after 1 year. A relative will also be interviewed once on postoperative day 13-16. Cognitive function will be measured preoperatively and on postoperative day 13-16 using the International Study Group of Postoperative Cognitive Dysfunction (ISPOCD) test battery. Symptoms / discomfort will be measured pre- and postoperatively (on postoperative day 1 and 2 and at the follow up visit day 13-16) by the Swedish version of Quality of Recovery (SwQoR) and by a visual analogue scale assessing pain intensity. Biomarkers will also be collected at the same time points. The findings from the interviews will be sorted out depending on group stratification (no delayed neurocognitive recovery and delayed neurocognitive recovery). The qualitative and quantitative findings will be compared to seek for similarities and differences.

DETAILED DESCRIPTION:
Aim The aim of present study is therefore to explore patients' experiences of their early and late postoperative cognition after major orthopaedic surgery in relation to postoperative cognitive function assessed with validated neuropsychological tests, inflammatory signalling molecules and quality of postoperative recovery as well as to describe the relative's view of early postoperative cognition.

Study design A mixed-methods study i.e. inductive concurrent design where, the core component is qualitative and the supplemental component is quantitative with integration of qualitative and quantitative data within a single investigation will be undertaken to address the research questions.

Participants Patients Participants included will be patients undergoing major elective joint replacement surgery (n=40) at a university hospital in Sweden. The sample size is based on the mixed methods study design and the incidence of early cognitive decline at 1-2 weeks postoperatively of 17% -25%.

Exclusion criteria: a score on the mini-mental state examination (MMSE) at screening of ≤ 22 i.e. suspected dementia; < 60 years of age; suffering from a nervous system disease; taking tranquillisers or antidepressants; underwent a surgical procedure in the previous six months; or inability to read and speak Swedish; suffering from a severe visual or auditory disorder, alcoholism or drug dependence.

Relatives One close relatives (spouses or children with age ≥ 18 years) per patients will be asked to participate. Inclusion criteria for the relatives included identifying themselves as being a relative whom the patient included in the study and being able to take part in an interview in Swedish. The patient decide which relative that should be asked. If the relative do not accept to be included, the patient will not be excluded.

Recruitment One of the researchers will, during their preoperative anaesthesia consultation, provide oral and written information about the study. The details of the study and its potential benefits as well as risks will be explained thoroughly to the patient. If the patient agrees to participation in the study, they will undergo the MMSE screening. Values >22 indicated that the patient is eligible to participate,

Qualitative data Interviews The patients and their relative will be interviewed separately. The opening question to the patients is: "How do you yourself experience the time after the operation compared to before? " Opening question to the relative: "How would you describe your relative regarding being as they used to be, being themselves, before the operation compared to the time after surgery" Probing questions were asked such as "What do you mean?" and "How would you describe that?" One year after the operation, a second interview with the patients will be conducted with a focus on their experiences of the postoperative recovery during the first year.

The informants will be encouraged to speak freely about the experience. An interview guide will be used to ensure covering issues such as cognition, memory loss, attention, mood and daily activity.

Quantitative data Cognitive Testing Cognitive function will be measured preoperatively and on postoperative day 13-16 using the International Study Group of Postoperative Cognitive Dysfunction (ISPOCD) neuropsychological test battery The ISPOCD battery assesses cognitive performance using four different tests, providing seven variables for analysis, including Visual Verbal Learning Test, the Concept Shifting Test, the Stroop Colour-Word Test, the Letter-Digit Coding Test 2 and has been validated in the perioperative setting for two decades. The tests will be administered in the same sequence at each test session by the same researcher following a standardized instruction manual in order to ensure as uniform a test situation as possible. The tests will be carried out in quiet rooms and only the patient and a researcher will be present.

Blood borne biomarkers Inflammatory signalling molecules such as CRP, Interleukin 1-beta, Interleukin-6, Interleukin-10, HMGB-1 and fractalkine will be measured preoperatively and postoperatively. Venous blood samples (20 mL whole blood) will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.

Quality of recovery The patients' quality of recovery will be measured with the Swedish Quality of Recovery (SwQoR), which measure 24 different items related to symptoms/discomfort that appear postoperatively, such as pain, anxiety, sleep difficulties, dizziness, fatigue, returning to work or usual home activities. The items are rated on 11-point numerical scales ranging from 0, "none of the time", to 10, "all of the time". Reliability and validity tests have provided evidence that it is appropriate to use SwQoR in patients undergoing surgery.

Pain intensity Pain intensity will be measured using a numerical rating scale (NRS) from 0 = no pain to 10 = maximum possible pain. The NRS has been tested for reliability and validity in a Swedish population26.

Demographic and perioperative data These include: age, sex, MMSE score, comorbidities, American Society of Anaesthesiologists classification, aesthetic technique and duration, duration of the procedure, blood loss (mL), blood transfusion (mL), use of analgesics during hospitalization and at home until the follow up visit, postoperative complications and length of stay.

Procedure Preoperative data collection If the patient chooses to participate in the study, they will undergo the cognitive test preoperatively. The test will be performed in an undisturbed room where only the patient and researchers will be present. The tests are expected to take about 20 minutes. Blood borne biomarkers will be collected and SwQoR and pain intensity questions will be measured after the cognitive testing is completed, The day and time of day for preoperative data collection will be documented.

Postoperative data collection The cognitive test and the interview with the patients will take place on postoperative day 13-16 during the patient's follow up visit. After the cognitive test is completed, SwQoR and biomarkers will be measured. The patient's relatives will be interviewed separately on the same day or the day after and by the same researcher . One year after the operation, a second interview with the patients will also be conducted. All cognitive tests will be performed by one of the researchers from the research group , with education and experience of performing the test. SwQoR, pain intensity and blood borne biomarkers will be measured postoperative day 1 to 3, the same time of day ±2 hours, and on day 13-16 during patient's follow up visit. The day and time of day for sampling biomarkers at the follow up visit will be documented. A research nurses at the Clinical Research Unit at the University Hospital will collect all biomarkers.

Data analysis Qualitative data analysis All interviews will be transcribed verbatim and analysed in line with an inductive thematic analysis . In the first step, all interviews will be read through, patients and relatives separately, and expressions concerning the experienced postoperative cognitive decline will be marked. At the same time, initial reflections on the data will be noted. In the second step, the marked expressions will be coded into a condensed, semantic description of the experiences expressed. Thirdly, themes will be identified, based on sorting the codes and initial reflections. In this step, relations between and levels of the themes will also be mapped. In step four, a review of the themes will be conducted, in which all codes included in a theme are considered, following which the whole analysis is considered in relation to the initial reflections and original texts. Thereafter, all themes and subthemes will be named. The findings from patients and relatives will be presented separately as well as being compared to seek for similarities and differences, and will be highlighted. Also, individual similarities and differences within the couples will be presented. The data analysis will be blinded to the findings from the biomarkers, cognitive tests, SwQoR and pain in order to not be influenced. The analysis will be performed in Swedish and thereafter be translated into English.

Quantitative data analysis Changes in cognitive performance will be calculated for each of seven test variables and corrected for practice effects and variability using data from a historical age-matched control group that has undergone testing using the same battery and with the same intervals2. To quantify the change from preoperative test to the postoperative tests scores, separate and composite Z-scores will be calculated on the basis of the seven cognitive test results and compared using Mann-Whitney U rank sum test.

To analyse differences in biomarkers within patients and between patients, Chi-square or student's t-tests will be used. To analyse differences within patients and between patients in cognitive performance and postoperative recovery, Mann-Whitney U rank sum tests will be used. For statistical analyses, IBM SPSS statistics version 24 for Windows will be used (IBM, Armonk, NY, USA). A p-value of <0.05 will be considered to be statistically significant in all analyses.

Descriptive statistics of demographic and perioperative data will be presented by number, percentage, and mean (SD) or min-max, as appropriate. Depending on the results from the cognitive tests and biomarkers, the patients will be stratified on the basis of their postoperative composite cognitive Z-score result into two groups; no delayed neurocognitive recovery corresponding to a composite Z-score <1 or delayed neurocognitive recovery with composite Z-score ≥ 1.0 2 Patient characteristics will be compared, between these two groups, using Fisher's exact test for categorical outcomes and t-tests or the Wilcoxon rank-sum test for continuous variables, as appropriate. A difference will be considered if any of these characteristics between the two groups has a p value of <0.05.

The analytical point of integration The qualitative and quantitative findings will be brought together to look for similarities i.e. whether the qualitative and the quantitative findings yields convergent results (triangulation) or if they are diverged. Thereafter the findings from the interviews, both patients and relatives will be sorted out depending on group stratification (no delayed neurocognitive recovery or delayed neurocognitive recovery). The qualitative and quantitative findings will then be compared to seek for similarities and differences. All patients will be included in the mixed data analysis even though they have an improvement in Z-score, SwQoR or biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* undergoing major elective joint replacement surgery

Exclusion Criteria:

* a score on the mini-mental state examination (MMSE) at screening of ≤ 22 i.e. suspected dementia
* age < 60 years
* suffering from a nervous system disease
* taking tranquillisers or antidepressants
* underwent a surgical procedure in the previous six months
* inability to read and speak Swedish
* suffering from a severe visual or auditory disorder, alcoholism or drug dependence

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major elective joint replacement surgery at a university hospital in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Patients experiences of early postoperative cognitive recovery | 13-16 days after surgery
  The opening question t: "How do you yourself experience the time after the operation compared to before? " Probing questions were asked such as "What do you mean?" and "How would you describe that?" The informants will be encouraged to speak freely about the experience. An interview guide will be used to ensure covering issues such as cognition, memory loss, attention, mood and daily activity.
Relatives experiences of patients early postoperative cognitive recovery | 13-16 days after surgery
  Opening question : "How would you describe your relative regarding being as they used to be, being themselves, before the operation compared to the time after surgery" Probing questions were asked such as "What do you mean?" and "How would you describe that?" The informants will be encouraged to speak freely about the experience. An interview guide will be used to ensure covering issues such as cognition, memory loss, attention, mood and daily activity.
Cognitive function | 13-16 days after surgery
  Cognitive function will be measured preoperatively and on postoperative day 13-16 using the International Study Group of Postoperative Cognitive Dysfunction (ISPOCD) neuropsychological test battery The ISPOCD battery assesses cognitive performance using four different tests, providing seven variables for analysis, including Visual Verbal Learning Test, the Concept Shifting Test, the Stroop Colour-Word Test, the Letter-Digit Coding Test and has been validated in the perioperative setting for two decades. The tests will be administered in the same sequence at each test session by the same researcher following a standardized instruction manual in order to ensure as uniform a test situation as possible. The tests will be carried out in quiet rooms and only the patient and a researcher will be present.
Quality of postoperative recovery | 13-16 days after surgery
  The patients' quality of recovery will be measured with the Swedish Quality of Recovery (SwQoR), which measure 24 different items related to symptoms/discomfort that appear postoperatively, such as pain, anxiety, sleep difficulties, dizziness, fatigue, returning to work or usual home activities. The items are rated on 11-point numerical scales ranging from 0, "none of the time", to 10, "all of the time". Reliability and validity tests have provided evidence that it is appropriate to use SwQoR in patients undergoing surgery

SECONDARY OUTCOMES:
Experiences of late postoperative cognitive recovery | 1 year after surgery
  One year after the operation, a second interview with the patients will be conducted with a focus on their experiences of the postoperative recovery during the first year. The informants will be encouraged to speak freely about the experience. An interview guide will be used to ensure covering issues such as cognition, memory loss, attention, mood and daily activity.
C-reactive protein (mg/L) | 13-16 days after surgery
  Venous blood samples. Measured preoperatively and postoperative day 1 and on day 13-16 during patient's follow up visit.enous blood samples will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.
Interleukin-6 (pg/mL) | 13-16 days after surgery
  Venous blood samples. Measured preoperatively and postoperative day 1 and on day 13-16 during patient's follow up visit.enous blood samples will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.
HMGB-1 (μg/mL) | 13-16 days after surgery
  Venous blood samples. Measured preoperatively and postoperative day 1 and on day 13-16 during patient's follow up visit.enous blood samples will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.
Interleukin 1-beta (pg/mL) | 13-16 days after surgery
  Venous blood samples. Measured preoperatively and postoperative day 1 and on day 13-16 during patient's follow up visit.enous blood samples will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.
Interleukin-10 (pg/mL) | 13-16 days after surgery
  Venous blood samples. Measured preoperatively and postoperative day 1 and on day 13-16 during patient's follow up visit.enous blood samples will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.
Fractalkine (pg/mL) | 13-16 days after surgery
  Venous blood samples. Measured preoperatively and postoperative day 1 and on day 13-16 during patient's follow up visit.enous blood samples will be drawn from an intravenous cannula. Blood will be centrifuged and plasma stored at -80 degrees C until further analysed.
Postoperative pain | 13-16 days after surgery
  Pain intensity will be measured using a numerical rating scale (NRS) from 0 = no pain to 10 = maximum possible pain. Postoperative pain intensity will be measured postoperative day 1 to 3, the same time of day ±2 hours, and on day 13-16 during patient's follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrica Nilsson, Principal Investigator — Karolinska Institutet
Locations (1):
- Ulrica Nilsson, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amirpour A, Bergman L, Markovic G, Liander K, Nilsson U, Eckerblad J. Understanding neurocognitive recovery in older adults after total hip arthroplasty-neurocognitive assessment, blood biomarkers and patient experiences: a mixed-methods study. BMJ Open. 2025 Jan 28;15(1):e093872. doi: 10.1136/bmjopen-2024-093872. PMID 39880425